CLINICAL TRIAL: NCT03638882
Title: Boosting Cognitive Reserve Through Adult Second Language Acquisition With Duolingo
Brief Title: Cognitive Reserve and Second Language Acquisition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Jed A. Meltzer, Ph.D, Neurorehabilitation Scientist, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: I2P2-2-00140
Record Dates: First submitted 2018-07-04; First posted 2018-08-20 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Executive Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Duolingo Spanish Course (Experimental): 30 minutes each day, 5 days a week for 16 weeks. Total of 40 hours.
  Interventions: Behavioral: Duolingo
- BrainHQ (Active Comparator): 30 minutes each day, 5 days a week for 16 weeks. Total of 40 hours.
  Interventions: Behavioral: BrainHQ
- Passive Control (Placebo Comparator): No intervention.
  Interventions: Behavioral: Passive Control

INTERVENTIONS:
Behavioral: Duolingo — Will learn Spanish using the commercially available Duolingo application. It is a computerized language training program.
  Arms: Duolingo Spanish Course
Behavioral: BrainHQ — Will use the commercially available Posit Science product Brain HQ. Brain HQ is a computerized adaptive cognitive brain training program.
  Arms: BrainHQ
Behavioral: Passive Control — No Intervention.
  Arms: Passive Control

SUMMARY:
Bilingualism has been shown to have a strong protective effect against dementia, delaying the diagnosis of Alzheimer's disease by up to 4 years. The purpose of the study is to test whether learning a second language using Duolingo software could improve cognitive functions in older adults.

DETAILED DESCRIPTION:
This study is a 3-arm, randomized controlled trial. The primary objective of the study is to test the impact of second language acquisition through short-term use of the Duolingo app on cognitive functioning, particularly executive function in older adults compared to a brain training application.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have normal vision and hearing.
* Participants must be able to travel to Baycrest by personal or study-arranged automobile, or public transportation.
* Participants must be monolingual native English speakers.
* Participants must be willing to provide informed consent.
* Participants must have daily access to a smartphone/mobile device.
* Have not previously studied Spanish formally, nor any other language in the past 10 years.

Exclusion Criteria:

* have a neurological disorder.
* meet DSM-IV-TR criteria for Axis I mood, anxiety, or psychotic or substance abuse disorders.
* Fluent in more than one language.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in working memory, n-back | change from baseline to 16 weeks
  Working memory assessed by the n-back test
Change in inhibitory Control, Simon task | change from baseline to 16 weeks
  Inhibitory control assessed by the Simon task
Change in inhibitory Control, DKEFS | change from baseline to 16 weeks
  DKEFS Colour Word Interference

SECONDARY OUTCOMES:
Change in attention abilities | change from baseline to 16 weeks
  Attention assessed by the Test of Everyday Attention (TEA)
Change in language abilities | change from baseline to 16 weeks
  Winterlight designed battery assessing paragraph reading and recall, picture description and object naming.
change in verbal fluency | change from baseline to 16 weeks
  semantic and phonological fluency tasks
executive function assessed by trailmaking test | change from baseline to 16 weeks
  Trails B implemented on tablet

OTHER OUTCOMES:
Spanish Proficiency (Duolingo group only) | change from baseline to 16 weeks
  WebCAPE Online Spanish Test

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada